CLINICAL TRIAL: NCT01085344
Title: Moderate Term Musculoskeletal Outcomes With Escalating Dose Prophylaxis: the Canadian Hemophilia Prophylaxis Study Follow-up Study
Brief Title: Canadian Hemophilia Prophylaxis Study
Acronym: CHPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian Feldman, Division Head, Rheumatology, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0019970022
Record Dates: First submitted 2010-03-01; First posted 2010-03-11 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Severe Hemophilia A
Keywords: hemophilia, prophylaxis, cost effectiveness
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Factor VIII (Experimental): escalating dose Factor VIII
  Interventions: Biological: Recombinant Factor VIII (Advate/Helixate FS/KoegenateFS)

INTERVENTIONS:
Biological: Recombinant Factor VIII (Advate/Helixate FS/KoegenateFS) — escalating dose prophylaxis
  Other Names: Recombinant Factor VIII (antihemophilic agent)
Biological: Recombinant Factor VIII (Advate/Helixate FS/KoegenateFS) — escalating dose
  Other Names: recombinant factor VIII (antihemophilic agent)

SUMMARY:
Primary prophylaxis given less frequently initially, with the infusion frequency increased if needed (Escalating Dose Prophylaxis), is likely to be less expensive and associated with fewer complications than standard prophylaxis while reducing disability to a greater degree than intermittent therapy.

DETAILED DESCRIPTION:
There are 2 specific study objectives. The first is to estimate the incidence of target joint bleeding in patients with severe hemophilia A treated (for primary prophylaxis) with Escalating Dose Prophylactic factor replacement. The second objective is to obtain accurate estimates of the direct and indirect costs associated with this protocol for use in a cost-effectiveness model (comparing Escalating Dose with standard prophylaxis and with intermittent therapy).

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A (factor level less than 2%).
* Age greater than 1 year and less than or equal to 2.5 years.
* Normal joints using the World Federation of Hemophilia orthopedic scale.
* Normal radiographs of joints in which bleeding has occurred using the World Federation of Hemophilia radiographic scale.
* Platelet count of > 150,000.
* Informed consent to participate.

Exclusion Criteria:

* Three or more clinically determined bleeds into any single elbow, knee or ankle.
* Presence or past history of a circulating inhibitor (level ≥ 0.5 Bethesda Units).
* Family judged to be non-compliant by the local hemophilia clinic director.
* Competing risk (symptomatic HIV infection, juvenile rheumatoid arthritis, metabolic bone disease, or other diseases known to cause or mimic arthritis.)

Ages: 12 Months to 30 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 1997-06-26 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Feldman, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Feldman BM, Rivard GE, Babyn P, Wu JKM, Steele M, Poon MC, Card RT, Israels SJ, Laferriere N, Gill K, Chan AK, Carcao M, Klaassen RJ, Cloutier S, Price VE, Dover S, Blanchette VS. Tailored frequency-escalated primary prophylaxis for severe haemophilia A: results of the 16-year Canadian Hemophilia Prophylaxis Study longitudinal cohort. Lancet Haematol. 2018 Jun;5(6):e252-e260. doi: 10.1016/S2352-3026(18)30048-6. Epub 2018 May 3. PMID 29731369

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 26, 1997, and Jan 30, 2007, 56 boys were enrolled from 12 Canadian centres.
Period: Overall Study
Arm/Group | Factor VIII
Started | 56
Completed | 50
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Factor VIII
Number analyzed (Participants) | 56
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 1.6 [1.2 to 2.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race or Ethnic Group: White European | 44
  Race or Ethnic Group: Mixed Aboriginal-Canadian | 5
  Race or Ethnic Group: Mixed Latin-American | 3
  Race or Ethnic Group: Asian | 2
  Race or Ethnic Group: African Heritage | 1
  Race or Ethnic Group: Middle Eastern | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed Target Joint Bleeding
Description: The number of participants who developed target joint bleeding during the study, which was defined as 3 bleeds into any 1 joint within a period of 3 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Factor VIII
Number analyzed (Participants) | 56
Participants | 17

2. Secondary Outcome: Annualized Bleeding Rate
Description: Number of index hemarthorses (bleeds into ankles, elbows or knees) per patient per year
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | Factor VIII
Number analyzed (Participants) | 56
episodes per participant per year | 0.95 [0.44 to 1.35]

3. Secondary Outcome: Annualized Factor Use
Description: annual factor usage per subject
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: IU/kg/year
Arm/Group | Factor VIII
Number analyzed (Participants) | 56
IU/kg/year | 3600 [3200 to 4700]

4. Secondary Outcome: Number of Patients Who Developed an Inhibitor to FVIII
Description: The number of patients who developed an inhibitor for FVIII, defined as >= 0.5 Bethesda Units
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Factor VIII
Number analyzed (Participants) | 56
Participants | 5

5. Secondary Outcome: Physical Disability as Measured by the CHAQ
Description: complete the Child Health Assessment Questionnaire (CHAQ) at each 6 month visit. The CHAQ is a validated tool to measure a disability index, with a possible score range of 0-3, where 0 represents no disability and 3 represents maximal disability. The CHAQ is known to have a strong ceiling effect.
  The CHAQ was collected at each study visit (i.e. every 6 months for the duration each patient was on study). The reported score represents the median end of study score.
Time Frame: through study completion, a median of 10 years
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Factor VIII
Number analyzed (Participants) | 56
units on a scale | 0 [0 to 0]

6. Secondary Outcome: Joint Damage as Determined by the Physiotherapy Score
Description: Complete the modified Colarado Physiotherapy Assessment every 6 months at each visit with a score range 0-30 for ankles and knees and 0-26 for elbows), measured at all study visits, which we modified by not assessing crepitus or the ankle joint circumference measurement. For each scale, 0 represents no joint damage, with 26/30 representing maximum possible joint damage. The reported score represents the median end of study score
Time Frame: through study completion, a median of 10 years
Population: Median CCPES Score at study-end
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Factor VIII
Number analyzed (Participants) | 56
units on a scale
  Left Ankle | 1 [0 to 12]
  Right Ankle | 1 [0 to 12]
  Left Elbow | 0 [0 to 7]
  Right Elbow | 0 [0 to 10]
  Left Knee | 0 [0 to 5]
  Right Knee | 0 [0 to 9]

7. Secondary Outcome: Complications Arising From Indwelling Venous Catheter
Description: collect information on any complications relating to indwelling venous catheters that some subject use.
Time Frame: 6 months
Population: 25 participants had a central venous access device (CVAD) during the study
Measure: Count of Participants; unit: Participants
Arm/Group | Factor VIII
Number analyzed (Participants) | 25
Participants | 0

ADVERSE EVENTS:
Arm/Group | Factor VIII
All-Cause Mortality (participants affected / at risk) | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No